CLINICAL TRIAL: NCT06420531
Title: A Multicenter Randomized Clinical Trial Comparing Two Human Milk Volumes to Optimize Growth and Gut Health in Infants Born Very Preterm
Brief Title: Milk And Growth In Children (MAGIC) Born Very Preterm: A Randomized Trial
Acronym: MAGIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013026
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Milk, Human

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: 180-200 mL/kg/day of human milk (Experimental): Study participants randomized to the intervention group will receive 180-200 mL/kg/day of human milk for 34 weeks corrected age.
  Interventions: Dietary Supplement: Human milk
- Control:140-160 mL/kg/day of human milk (Placebo Comparator): Study participants randomized to the control group will receive 140-160 mL/kg/day of human milk for 34 weeks corrected age.
  Interventions: Dietary Supplement: Human milk

INTERVENTIONS:
Dietary Supplement: Human milk — maternal breastmilk or donor breastmilk

SUMMARY:
The goal of this multi-center randomized, parallel group trial is to determine the effect of human milk diets ranging between 180 and 200 mL/kg/day on the body composition outcomes of moderately preterm infants born between 27 and 31 weeks of gestation.

DETAILED DESCRIPTION:
Participants will be randomized once they reach 120 mL/kg/day. Clinicians will be able to increase feeds each day as they see fit, until the patient reaches the target goal of 140-160 mL/kg/day or 180-200 mL/kg/day. They will then maintain this volume until 34 weeks postmenstrual age. Researchers will compare these two targets to see if higher feeding volumes prevent faltering growth without causing adverse metabolic outcomes.

Participants will:

* Have a feeding volume of 180-200 mL/kg/day or a volume of 140-160 mL/kg/day until 34 weeks corrected age
* Have four body composition assessments with a bioelectrical impedance analyzer throughout study period
* Have four stool samples collected throughout study period
* Have four maternal breastmilk samples collected and analyzed throughout the study period
* Have one blood sample collected at 36 weeks corrected age
* Have the option to participate in a follow-up survey completed by parents at 2-3 years of age

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 27 0/7 and 31 6/7 weeks
* Birthweight of 1500 grams or less
* Human milk feeding during the first 14 days after birth
* Full enteral feeding (120mL/kg/day or more) within the first 14 days after birth

Exclusion Criteria:

* Necrotizing enterocolitis stage 2 or greater
* Spontaneous intestinal perforation
* Major congenital/chromosomal anomalies
* Terminal illness requiring limited or withheld support
* Intention to restrict fluid intake after the first 14 postnatal days due to the presence of a symptomatic patent ductus arteriosus (PDA)
* Any formula feeding within the first 14 days after birth

Ages: 6 Hours to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 486 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Fat-free Mass (FFM)-For-age-Z-score | 36 weeks post menstrual age or hospital discharge, up to 120 days following birth, whichever is longer
  Estimated by bioelectric impedance analysis. FFM measurements will be converted into Z-scores using updated, sex specific reference curves of body composition in preterm infants

SECONDARY OUTCOMES:
Body fat percentage | Birth to 36 weeks postmenstrual age
  Estimated by bioelectric impedance analysis. Body fat measurements will be converted into Z-scores using updated sex-specific reference curves of body composition in preterm infants.
Anthropometric Measurements | Birth to 36 weeks postmenstrual age
  Weight, length, head circumference, and mid-upper arm circumference measurements. Measurements will be converted into Z-scores based on Fenton growth curves (2013).
Bronchopulmonary Dysplasia | 36 weeks post menstrual age or hospital discharge, up to 120 days following birth, whichever is longer
  Number of participants receiving supplemental oxygen at 36 weeks (PMA)
Number of Days Alive and Receiving Full Enteral Feeding | Birth to 28 days
  Time to full enteral feeding days
Duration of Hospital Stay in Days | Birth to 120 days or discharge, whichever occurs first
  From day of admission to day of hospital discharge to home
Growth Rate | Birth to 36 weeks postmenstrual age or hospital discharge (whichever occurs first).
  Weight gain in g/kg/day
Number of Participants with Postnatal Faltering Growth | 36 weeks or hospital discharge (whichever occurs first)
  Diagnosis of faltering growth (weight z score decline from birth to 36 weeks > 1) using the 2013 Fenton growth curve.
Number of Participants diagnosed with Necrotizing Enterocolitis | From birth up to 120 days following birth
  Diagnosis of necrotizing enterocolitis stage 2 or 3
Number of Participants with Diagnosis of Intestinal Perforation | From birth up to 120 days following birth
  Diagnosis of intestinal perforation
Death | Birth to 120 days
  Death prior to 121 days of life
Culture-proven Sepsis | Birth to 120 days
  Diagnosis of sepsis with positive blood cultures
Fat Mass (FM)- For age Z-score | 36 weeks or hospital discharge, up to 120 days following birth, whichever is longer
  Estimated by bioelectric impedance analysis. FM measurements will be converted into Z-scores using updated sex-specific reference curves of body composition in preterm infants.
Body Fat (BF)-For age Z-score | 36 weeks post menstrual age or hospital discharge, up to 120 days following birth, whichever is longer
  Estimated by bioelectric impedance analysis. BF measurements will be converted into Z-scores using updated sex-specific reference curves of body composition in preterm infants.
Duration of parenteral nutrition | Birth to 28 days of life
  Number of days receiving parenteral nutrition
Post discharge growth outcomes | 22-26 months corrected age
  Weight, length, and head circumference measurements. Measurements will be converted into Z-scores.

OTHER OUTCOMES:
Changes in Intestinal Microbiome | Birth to 36 weeks postmenstrual age
  Determined by molecular analyses of fecal samples
Changes in Metabolic Pathways | 36 weeks postmenstrual age or discharge (whichever occurs first)
  Determined by molecular analyses of serum samples
Cognitive scores | 2 - 3 years of age
  Neurodevelopmental outcomes measured by voluntary PARCA-R survey

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — UAB Hospital
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas